CLINICAL TRIAL: NCT02708953
Title: Thoracic Spine Thrust Manipulation for Cervicogenic Headaches: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15-0983
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Headache Disorders, Secondary
MeSH Terms: conditions — Headache Disorders, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (thoracic manipulation) (Experimental): Patients in the initial manipulation group will attend physical therapy two sessions per week for 3 weeks for a total of 6 sessions. Each treatment session will last for a total of 15 minutes. After the initial manipulation group receives 3 weeks of treatment they will wait for 1-week, be retested, and then crossover into the other group.
  Interventions: Procedure: Thoracic manipulation (Manipulation Group)
- Wait-list (thoracic manipulation) (Active Comparator): When individuals are assigned to the wait-list control group they will serve as the control for 3 weeks while the initial manipulation group receives treatment. After serving as the wait-list control condition for 3 weeks, this group will then return for testing and will receive the manipulation package as described below at 4 weeks.
  Interventions: Procedure: Thoracic Manipulation (Control wait-list)

INTERVENTIONS:
Procedure: Thoracic manipulation (Manipulation Group) — Manipulation techniques will include: CT junction manipulation seated and supine, upper thoracic manipulation, middle thoracic spine manipulation in seated and supine, middle thoracic spine manipulation in prone, thoracic active range of motion exercise and instruction to maintain usual activity level within the limits of pain.
  Other Names: Manual therapy to thoracic spine
  Arms: Treatment (thoracic manipulation)
Procedure: Thoracic Manipulation (Control wait-list) — Manipulation techniques will include: CT junction manipulation seated and supine, upper thoracic manipulation, middle thoracic spine manipulation in seated and supine, middle thoracic spine manipulation in prone, thoracic active range of motion exercise and instruction to maintain usual activity level within the limits of pain.
  Other Names: Manual therapy to thoracic spine
  Arms: Wait-list (thoracic manipulation)

SUMMARY:
Headaches have been listed as 1 of the 10 most disabling conditions worldwide. (Stovner et al., 2007) and cervicogenic headaches (CeHs) comprise 15% of the individuals with these complaints. (Nillsson, 1995); (Fernandez de-las-penas et al., 2005) The current best approach to the conservative care of this condition has yet to be determined. The primary aim of this study is to determine whether individuals with CeHs will respond to a program of thoracic spine thrust manipulation in isolation. This may further the current body of evidence by offering an alternative, potentially safer approach to the conservative care of individuals with this condition. Additionally, results of this study may serve to drive a larger scale Randomized Clinical Trial (RCT) by offering information regarding feasibility of recruitment of individuals with chronic CeHs as well as timing and dosing of the intervention.

DETAILED DESCRIPTION:
Headaches have been listed as 1 of the 10 most disabling conditions worldwide. (Stovner et al., 2007) and cervicogenic headaches (CeHs) comprise 15% of the individuals with these complaints. (Nillsson, 1995); (Fernandez de-las-penas et al., 2005) The current best approach to the conservative care of this condition has yet to be determined. Evidence suggests that manipulative therapy aimed at the cervical spine in combination with exercise is helpful in alleviating these symptoms. (Jull et al., 2002) The risk of injury from cervical spine manipulative techniques has been documented to be remote (Haldeman et al., 2002; DiFabio 1999), however the potential consequences can be severe. Therefore with inherently lower risks, thoracic spine manipulations may be a suitable alternative as the evidence is accumulating for its influence on the cervical spine. (Mintken et al., 2010; Boyles et al., 2009; Cleland et al., 2005 & 2007 A & B, 2010; Flynn et al., 2001; Fernandez-de-las-penas et al., 2004; Piva et al., 2000; Browder et al., 2004) The primary aim of this study is to determine whether individuals with CeHs will respond to a program of thoracic spine thrust manipulation in isolation. This may further the current body of evidence by offering an alternative, potentially safer approach to the conservative care of individuals with this condition. Additionally, results of this study may serve to drive a larger scale RCT by offering information regarding feasibility of recruitment of individuals with chronic CeHs as well as timing and dosing of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 60 years old Sjaastad et al for CeH, which included
* unilateral or unilateral dominant side-consistent headache associated with neck pain and aggravated by neck postures or movement (Sjaastad et al., 1998)
* joint tenderness in at least one of the three upper cervical joints (C0-C3) as assessed by manual palpation
* headache frequency of at least one per week over the past 2 months

Exclusion Criteria:

* red flags noted in the patient's Neck Medical Screening Questionnaire (e.g. tumor, fracture)
* metabolic diseases RA, osteoporosis, prolonged history of steroid use, symptoms of vertebrobasilary insufficiency, pregnancy, cervical spinal stenosis, bilateral upper extremity symptoms etc.)
* history of whiplash injury within the past six weeks
* evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes
* two or more positive neurologic signs consistent with nerve root compression, including any two of the following: muscle weakness involving a major muscle group of the upper extremity, diminished upper extremity muscle stretch reflex (biceps brachii, brachioradialis, or triceps reflex), diminished or absent sensation to pinprick in any upper extremity dermatome
* prior surgery to the neck or thoracic spine
* chiropractic or physical therapy treatment for their headaches over the past 6-months
* bilateral headache description
* migraine headaches with or without aura
* workers compensation or pending legal action regarding their headaches
* inability to comply with treatment and follow-up schedule
* we will not recruit individuals whom the researcher is in a position to punish or reward, whether through grades, evaluations, or promotions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Headache Disability Index | Baseline
  Headache Disability Index (HDI): The HDI is a 25-item questionnaire used to assess the patient's perceived impact of the headaches on their daily life.
Headache Disability Index | 4 weeks
  Headache Disability Index (HDI): The HDI is a 25-item questionnaire used to assess the patient's perceived impact of the headaches on their daily life.
Headache Disability Index | 8 weeks
  Headache Disability Index (HDI): The HDI is a 25-item questionnaire used to assess the patient's perceived impact of the headaches on their daily life.
Headache Disability Index | 3 months
  Headache Disability Index (HDI): The HDI is a 25-item questionnaire used to assess the patient's perceived impact of the headaches on their daily life.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | Baseline
  An 11-point NPRS will be used to measure pain intensity. Patients rate their current level of pain and their worse and least amount of pain in the last 24 hours.
Numeric Pain Rating Scale | 4 weeks
  An 11-point NPRS will be used to measure pain intensity. Patients rate their current level of pain and their worse and least amount of pain in the last 24 hours.
Numeric Pain Rating Scale | 8 weeks
  An 11-point NPRS will be used to measure pain intensity. Patients rate their current level of pain and their worse and least amount of pain in the last 24 hours.
Numeric Pain Rating Scale | 3 months
  An 11-point NPRS will be used to measure pain intensity. Patients rate their current level of pain and their worse and least amount of pain in the last 24 hours.
Pain Self Efficacy Questionnaire (PSEQ) | Baseline
  The 10 item questionnaire is used to assess the patient's confidence in performing specific activities despite pain. Items are listed on a 0 to 6 scale, with a maximum score of 60 points.
Pain Self Efficacy Questionnaire (PSEQ) | 4 weeks
  The 10 item questionnaire is used to assess the patient's confidence in performing specific activities despite pain. Items are listed on a 0 to 6 scale, with a maximum score of 60 points.
Pain Self Efficacy Questionnaire (PSEQ) | 8 weeks
  The 10 item questionnaire is used to assess the patient's confidence in performing specific activities despite pain. Items are listed on a 0 to 6 scale, with a maximum score of 60 points.
Pain Self Efficacy Questionnaire (PSEQ) | 3 months
  The 10 item questionnaire is used to assess the patient's confidence in performing specific activities despite pain. Items are listed on a 0 to 6 scale, with a maximum score of 60 points.

CONTACTS AND LOCATIONS:
Overall Officials: Amy W McDevitt, DPT, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jull G, Trott P, Potter H, Zito G, Niere K, Shirley D, Emberson J, Marschner I, Richardson C. A randomized controlled trial of exercise and manipulative therapy for cervicogenic headache. Spine (Phila Pa 1976). 2002 Sep 1;27(17):1835-43; discussion 1843. doi: 10.1097/00007632-200209010-00004. PMID 12221344